CLINICAL TRIAL: NCT05855382
Title: A Prevalence Study of Persistent COVID-19 in Punta Arenas, Magallanes and Chilean Antarctic Region
Brief Title: Prevalence of Persistent COVID-19 in Punta Arenas, Magallanes and Chilean Antarctic Region
Acronym: PCOV-19
Status: Recruiting | Type: Observational
Sponsor: Universidad de Magallanes (Other)
Collaborators: Centro Asistencial Docente e Investigación de la Universidad Magallanes (CADI-UMAG) (Unknown); University of Chile (Other); Universidad de Santiago de Chile (Other)
Responsible Party: Principal Investigator, Marcelo A. Navarrete Signorile, Principal Investigator, Universidad de Magallanes
Other Study IDs: FIC-R 40036196-0
Record Dates: First submitted 2023-05-07; First posted 2023-05-11 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 13 Months
Biospecimen Retention: Samples With DNA — * Full blood count: red cell count, haemoglobin, haematocrit, mean cellular volume (MCV), mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), red cell distribution width (RDW), white cell count and differential (neutrophil count, lymphocyte count, monocyte count, eosinophil count, and basophil count), and platelet count.
  * Biochemical profile: Urea/urea nitrogen, Creatinine, Total protein, Albumin,Total bilirubin, Alkaline phosphatase (ALP),Transaminases GOT/GPT, Uric acid, Total cholesterol, Triglycerides, Glucose, Calcium, Phosphorus.
  * Vitamin D.
  * Blood sample molecular analysis: inflammatory biomarkers(IL-8, IL-1β, IL-6, IL-10, TNF e IL-12p70), lymphocyte subpopulations, Age-associated B cells (ABCs), Immunological repertoire.
  * DNA extraction for genotyping and sequencing at the Centro Austral de Tecnología Genómica (cATG).
  * Additional peripheral blood mononuclear cell (PBMC) and serum samples will be stored for possible future analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Adults with at least one positive SARS-CoV-2 RT-qPCR test
  Interventions: Other: Persistent COVID-19

INTERVENTIONS:
Other: Persistent COVID-19 — To determine the prevalence of persistent COVID-19 diagnosis in the current study, we will identify adults between 18 and 100 years of age who have had at least one positive SARS-CoV-2 RT-qPCR test from the COVID-19 database maintained by the SEREMI of Health in Punta Arenas between July 2022 and July 2023.

SUMMARY:
This cross-sectional observational study aims to determine the prevalence of Persistent COVID-19 in 282 individuals in Punta Arenas, Magallanes and Chilean Antarctic Region. Persistent COVID-19 is a complex array of symptoms that persist or emerge for more than 4 weeks beyond SARS-CoV-2 infection. Recent studies suggest that up to 80% of survivors may develop chronic multi-organ dysfunction due to persistent inflammation and immune dysregulation, making it an ongoing public health concern worldwide.

The study aims to (1) describe and establish the frequency of physical and psychological signs and symptoms in adult patients who have tested positive for COVID-19, (2) identify individuals who meet the WHO case definition of Persistent COVID-19 in Chile, (3) explore risk factors associated with persistent COVID-19 to guide intervention strategies, and (4) explore inflammatory and molecular biomarkers associated with persistent COVID-19.

The research project utilizes a stratified random sampling with a mixed-methods embedded design. In the first phase, individuals diagnosed with COVID-19 will be recruited and followed up to complete the study's sample universe. A sociodemographic survey, blood sampling (including complete blood count, biochemical profile, immunoglobulin mutational status analysis, and analysis of inflammatory biomarkers), and a battery of psychological tests will be administered. In the second phase, kinesiology studies and medical consultation and evaluation will be conducted to determine if individuals have Persistent COVID-19 and to derive them to the healthcare network. In the final follow-up phase, participants diagnosed with Persistent COVID-19 will be invited to undergo musculoskeletal and respiratory assessments to complete the diagnosis of symptoms associated with the pathology.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Individuals must be included in the COVID-19 monitoring database by the SEREMI of Health in Punta Arenas between July 2022 and July 2023.
* Patients able to give informed consent.

Exclusion Criteria:

* Age < 18 years
* Any physical, mental, immunosuppressive, or social condition that, in the investigator's judgment, might interfere with the completion of the baseline assessments and evaluations.
* Individuals who are digitally illiterate and do not have access to nearby networks to support them during the process.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To identify potential participants for this population-based study with stratified random sampling, we also considered the following eligibility criteria: (1) Diagnosed SARS-CoV-2 infection confirmed by RT-qPCR test (2) residency in Punta Arenas, (3) recruitment messages via phone calls, text messages, emails, and social media postings, and (4) referrals from collaborating healthcare providers.
Sampling Method: Probability Sample
Enrollment: 282 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
To determine the prevalence of persistent COVID-19 in a cohort of patients in Punta Arenas | 13 months

SECONDARY OUTCOMES:
Sociodemographic data questionnaire | 3 months
  to determine the number of prior illnesses, medical treatments, and vaccination records, as well as the quality of life scales, persistent COVID-19 symptoms through self-reported survey data, and Informed Consent Comprehension Questionnaire.
Psychological profiles | 3 months
  Beck Anxiety Scale (BAI)
Psychological profiles | 3 months
  D2-R test of attention
Psychological profiles | 3 months
  Wechsler Adult Intelligence Scale (WAIS)
Sleep quality and disorders | 3 months
  Pittsburgh Sleep Quality Index (PSQI)
Psychosocial exposures | 3 months
  COVID-19 related stress questionnaire based on the Perceived Stress Scale
Psychosocial exposures | 3 months
  Normal activities and work productivity questionnaire; daily diaries
Standard laboratory parameters | 3 months
  Full blood count
Standard laboratory parameters | 3 months
  Serum chemistry test
Inflammatory Biomarkers | 6 months
  Interleukin-8 (IL-8)
Inflammatory Biomarkers | 6 months
  Interleukin-1β (IL-1β)
Inflammatory Biomarkers | 6 months
  Interleukin-6 (IL-6)
Inflammatory Biomarkers | 6 months
  Interleukin-10 (IL-10)
Inflammatory Biomarkers | 6 months
  Tumor Necrosis Factor (TNF)
Inflammatory Biomarkers | 6 months
  Interleukin-12 (IL-12p70)
Immunological repertoire associated with persistent COVID-19 | 6 months
  DNA sequencing results
Flow Cytometry Immunophenotyping | 6 months
  Quantify different lymphocyte subpopulations in persistent COVID-19
Flow Cytometry Immunophenotyping | 6 months
  Quantify Age-Associated B Cells and Their Potential Role in Persistent COVID-19 Pathogenesis
Function of the musculoskeletal system | 6 months
  Fatigue Assessment Scale (FAS)
Function of the musculoskeletal system | 6 months
  Body Composition Analysis Assessment
Function of the musculoskeletal system | 6 months
  Hand Grip Strength Test
Function of the musculoskeletal system | 6 months
  Maximum inspiratory pressure test (MIP test)
Diagnosis of prevalent COVID-19 | 8 months
  Clinical determination of whether the patient has persistent COVID-19 or not is necessary for referral to the appropriate healthcare system

OTHER OUTCOMES:
Musculoskeletal Capacity | 2 months
  Heart Rate Variability (HRV) analysis
Musculoskeletal Capacity | 2 months
  walk test (distance): 3D temporal scanning system for gait analysis by photogrammetry
Musculoskeletal Capacity | 2 months
  Postural Stability and Control Assessment Using Balance Tests
Respiratory function: | 2 months
  Spirometry: measurement of respiratory flows and volumes.

CONTACTS AND LOCATIONS:
Locations (1):
- Teaching and Research Healthcare Center of the University of Magallanes (CADI-UMAG), Punta Arenas, Magllanes and Chilean Antartic Region, Chile

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared is all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following our data is cleaned, quality checked, and analyzed, we will make the data available to the general research community. All data made available for public use will be de-identified data, i.e., stripped of private, protected health information that could be used to deduce the identity of individual subjects, in compliance with the Rule.
Access Criteria: PPCov-19 Study website to be determined

REFERENCES:
- [Result] Gonzalez-Puelma J, Aldridge J, Montes de Oca M, Pinto M, Uribe-Paredes R, Fernandez-Goycoolea J, Alvarez-Saravia D, Alvarez H, Encina G, Weitzel T, Munoz R, Olivera-Nappa A, Pantano S, Navarrete MA. Mutation in a SARS-CoV-2 Haplotype from Sub-Antarctic Chile Reveals New Insights into the Spike's Dynamics. Viruses. 2021 May 11;13(5):883. doi: 10.3390/v13050883. PMID 34064904
- [Result] Sarmiento Varon L, Gonzalez-Puelma J, Medina-Ortiz D, Aldridge J, Alvarez-Saravia D, Uribe-Paredes R, Navarrete MA. The role of machine learning in health policies during the COVID-19 pandemic and in long COVID management. Front Public Health. 2023 Apr 11;11:1140353. doi: 10.3389/fpubh.2023.1140353. eCollection 2023. PMID 37113165
- [Result] Alvarado-Aravena C, Arriaza K, Castillo-Aguilar M, Flores K, Dagnino-Subiabre A, Estrada-Goic C, Nunez-Espinosa C. Effect of Confinement on Anxiety Symptoms and Sleep Quality during the COVID-19 Pandemic. Behav Sci (Basel). 2022 Oct 17;12(10):398. doi: 10.3390/bs12100398. PMID 36285967
- [Derived] Sarmiento Varon L, Alvarez H, Huirimilla Casanova LC, Diaz Mora MP, Munoz Cuevas LA, Gonzalez-Puelma J, Espinoza K, Amarales L, Luhr Henriquez J, Retamal-Matus F, Uribe-Paredes R, Nunez-Espinosa CA, Estrada-Goic C, Bachelet VC, Lopez Nitsche MN, Navarrete MA. Estimating the prevalence of persistent symptoms after SARS-CoV-2 infection (post-COVID-19 syndrome): a regional cross-sectional study protocol. BMJ Open. 2025 May 30;15(5):e093844. doi: 10.1136/bmjopen-2024-093844. PMID 40447416
- See also: Enrolling for the study — https://redcap.catg.cl/surveys/?s=9D4CRJYC4MNXTRA8